CLINICAL TRIAL: NCT02529813
Title: CD19+ Chimeric Antigen Receptor T Cells for Patients With Advanced Lymphoid Malignancies
Brief Title: CD19-Specific T-cells in Treating Patients With Advanced Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ziopharm Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1018; NCI-2015-01492 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20152145; 1159157; 2013-1018 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia; Blasts 5 Percent or More of Bone Marrow Nucleated Cells; CD19 Positive; Minimal Residual Disease; Non-Hodgkin Lymphoma; Small Lymphocytic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine phosphate; tisagenlecleucel; CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm I (CD19 positive chimeric antigen receptor T-cells) (Experimental): LYMPHODEPLETING CHEMOTHERAPY: Patients may receive standard chemotherapy comprised of fludarabine phosphate IV over 1 hour and cyclophosphamide IV over 3 hours on days -5 to -3 or cyclophosphamide IV every 12 hours on days -5 to -3 at the discretion of the treating physician.
  Within 30 days post completion of lymphodepletion, patients receive CD19 positive chimeric antigen receptor T-cells IV over 15-30 minutes on day 0, or split into two portions on days 0 and 1.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Tisagenlecleucel

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Tisagenlecleucel — Given IV
  Other Names: CART-19; CART19; CTL019; CTL019 T-cells; Kymriah; Tisagenlecleucel-T

SUMMARY:
This phase I clinical trial studies the side effects and best dose of CD19-specific T-cells in treating patients with lymphoid malignancies that have spread to other places in the body and usually cannot be cured or controlled with treatment. Sometimes researchers change the deoxyribonucleic acid (DNA) (genetic material in cells) of donated T-cells (white blood cells that support the immune system) using a process called "gene transfer." Gene transfer involves drawing blood from the patient, and then separating out the T-cells using a machine. Researchers then perform a gene transfer to change the T-cells' DNA, and then inject the changed T-cells into the body of the patient. Injecting modified T-cells made from the patient may help attack cancer cells in patients with advanced B-cell lymphoma or leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerated dose of genetically modified, CD19-specific T cells administered into patients with CD19+ advanced lymphoid malignancies.

SECONDARY OBJECTIVES:

I. To screen for the development of host immune responses against the CD19-specific chimeric antigen receptor (CAR).

II. To describe the homing ability of the infused T cells. III. To assess disease response. IV. To determine persistence of CAR+ T cells.

OUTLINE: This is a dose escalation study of CD19 positive chimeric antigen receptor T-cells.

LYMPHODEPLETING CHEMOTHERAPY: Patients may receive standard chemotherapy comprised of fludarabine phosphate intravenously (IV) over 1 hour and cyclophosphamide IV over 3 hours on days -5 to -3 or cyclophosphamide IV every 12 hours on days -5 to -3 at the discretion of the treating physician.

Within 30 days post completion of lymphodepletion, patients receive CD19 positive chimeric antigen receptor T-cells IV over 15-30 minutes on day 0, or split into two portions on days 0 and 1.

After completion of study treatment, patients are followed up for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of CD19+ lymphoid malignancy defined as acute lymphoblastic leukemia, acute biphenotypic leukemia, non-Hodgkin's lymphoma, small lymphocytic lymphoma, or chronic lymphocytic leukemia with active disease defined by presence of > 5% malignant blasts in bone marrow and/or peripheral blood, and/or minimal residual disease by flow cytometry or molecular analysis for fusion proteins, and/or positive imaging for extramedullary disease; patients must have measurable disease at time of study treatment
* Confirmed history of CD19 positivity by flow cytometry for malignant cells
* Lansky/Karnofsky performance scale > 60%
* Patient able to provide written informed consent; parent or guardian of minor patient able to provide written informed consent
* Patient able to provide written informed consent for the long-term follow-up gene therapy study: 2006-0676; parent or guardian of minor patient able to provide written informed consent for the long-term follow-up gene therapy study: 2006-0676

Exclusion Criteria:

* Positive beta human chorionic gonadotropin (HCG) in female of child-bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization or lactating females
* Patients with known allergy to bovine or murine products
* Positive serology for human immunodeficiency virus (HIV)
* Active hepatitis B or active hepatitis C
* Has received donor lymphocyte infusion (DLI) product within 6 weeks of CAR T cell infusion
* Has received allogeneic hematopoietic stem cell transplant within 3 months of CAR T cell infusion; hematopoietic stem cell transplant (HSCT) > 3 months from CAR T cell infusion eligible

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of genetically modified, CD19-specified T cells | Up to 30 days
  Will be defined as the highest dose for which the posterior probability of toxicity is closest to 25%. Demographic and clinical characteristics will be summarized using descriptive statistics by dose level. The number of patients with dose limiting toxicities will be reported at each dose level.

SECONDARY OUTCOMES:
The proportion of patients for which a T cell product could not be prepared | Up to 1 year
  Computed with a corresponding 95% confidence interval.
Proportion of patients experiencing response (complete response and partial response) | Up to 1 year
  Estimated with a corresponding 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org